CLINICAL TRIAL: NCT04932421
Title: Emotion Detectives - Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Children: A Randomized Controlled Trial in the Portuguese Population
Brief Title: Unified Protocol for Children: A Randomized Controlled Trial for the Portuguese Population
Acronym: UP-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Centro Hospitalar Tondela-Viseu (Other)
Responsible Party: Principal Investigator, Brigida Caiado, Dra. , PhD student, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Univeristy of Coimbra
Record Dates: First submitted 2021-05-31; First posted 2021-06-21 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Anxiety Disorders; Mood Disorders; Emotional Disorder; Emotional; Disorder, Childhood, With Anxiety and Fearfulness; Child Mental Disorder; Parenting
Keywords: emotional disorders; anxiety and mood disorders; children; parenting; transdiagnostic; unified protocol; randomized controlled trial
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: 1. experimental group (i.e., children and parents who benefit from the UP-C program).
  2. control group (i.e., children who benefit from a psychoeducational intervention program, named "ABC of Emotions").
Who Masked: Investigator
Masking Description: Single-blind - the investigator is unaware of the intervention assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (UP-C intervention) (Experimental): UP-C intervention 15 weekly sessions, for children and parents
  Interventions: Behavioral: Emotion Detectives: Unified protocol for transdiagnostic treatment of emotional disorders in children (UP-C)
- Control group (ABC of emotions intervention) (Active Comparator): ABC of emotions - a psychoeducational intervention 5 sessions every 3 weeks for children
  Interventions: Other: ABC of Emotions

INTERVENTIONS:
Behavioral: Emotion Detectives: Unified protocol for transdiagnostic treatment of emotional disorders in children (UP-C) — UP-C is a transdiagnostic and emotion-focused cognitive-behavioral group intervention for children aged 6-13 years old with emotions disorders (i.e., anxious and/or mood disorders) and their parents. UP-C unifies cognitive-behavioral, contextual (eg. mindfulness) and parental training techniques aiming to reduce the intensity and frequency of children's clinical symptomatology.
  The intervention consists of 15 weekly group sessions (90 minutes per session; 5-8 children and parents per group) conducted by at least two clinical psychologists trained in the UP-C. The sessions start with the parents and children together (15 minutes); then, one psychologist conduct the session with the group of children while the other psychologist conduct the session with the group of parents, simultaneously (60 minutes); finally, the session ends with the group together (15 minutes). This is a structured and manualized intervention with a manual for the therapist and a workbook for the child and parents.
  Other Names: UP-C
  Arms: Experimental group (UP-C intervention)
Other: ABC of Emotions — ABC of Emotions is a psychoeducational group intervention for children with anxiety and/or mood disorders, aged between 6 to 13 years. ABC of Emotions consists of 5 group psychoeducation sessions (about 90 minutes per session; 5-8 children per group). This is a structured and manualized intervention, with a manual for the therapist and a workbook for the child.
  The contents of the sessions were developed by the researchers of this study and are based on classic psychoeducational cognitive-behavioral therapies (CBT) strategies. Since anxiety disorders are more frequent in childhood than mood disorders (e.g., Merikangas et al., 2009), this program is essentially based on psychoeducation materials focused on emotions such as anxiety and fear. However, the same materials are available in an attachment, adapted for use with children to whom the main emotion is not fear/anxiety, but sadness (as in mood disorders).
  Arms: Control group (ABC of emotions intervention)

SUMMARY:
The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Children (UP-C) is a transdiagnostic and emotion-focused cognitive-behavioral group intervention for children aged 6-12 years old with emotion disorders (i.e., anxious and/or mood disorders) and their parents.

UP-C consists of 15 weekly group sessions and unifies cognitive-behavioral, contextual (e.g., mindfulness) and parental training techniques, for parents and children, aimed at reducing the intensity and frequency of strong and aversive emotional experiences in children and their clinical symptomatology.

The present study aims to assess the feasibility, acceptability and efficacy of the UP-C in the Portuguese population in reducing children's anxiety/depression symptoms. It also aims to investigate which mechanisms explain the therapeutic change.

Participants will be recruited at child mental health services and schools from Central Portugal and also through online dissemination of the study.

A randomized controlled trial (RCT) will be conducted in a sample of children aged 6-13 years old with emotional disorders and their parents in order to answer the critical question of whether the UP-C is more efficacious in reducing children's symptomatology than a psychoeducational group intervention (active control group).

Once the eligibility criteria are met (assessed by the project researchers) parents and children will be randomly assigned to one of two study conditions:

1. experimental group (i.e., children and parents who benefit from the UP-C program).
2. control group (i.e., children who benefit from a psychoeducational intervention program, named "ABC of Emotions").

Parents and children from both groups will complete several psychometrically robust and developmentally appropriate measures at baseline (T0), mid-treatment (only at week 7 of the UP-C; T1), post treatment (T2) and at 3 months follow-up (T3).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-13
* Primary diagnosis of an anxiety and/or depression disorder
* Speaking, reading and understanding Portuguese

Exclusion Criteria:

* Diagnosis of a psychotic disorder, bipolar disorder or intellectual disability;
* Severe current suicidal/homicidal ideation;
* The child is not on a stable dose of a psychotropic or other type of medication for at least 1 month prior to T0 assessment.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Changes of children's anxiety and depression | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
Changes of children's severity of psychopathology and improvement | Baseline, Póst treatment (15 weeks)
  Measured with an adaptation of Clinical Global Impression (CGI). The CGI is composed by a severity of illness scale and a scale evaluating changes from the initiation of treatment. Higher scores are indicative of higher severity of psychopathology and lower improvement from the initiation of treatment.

SECONDARY OUTCOMES:
Changes of child anxiety life interference | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Child Anxiety Life Interference Scale - self-report (CALIS-C) and parent's report (CALIS-P). The child form is composed by a single scale and the parent form is composed by two subscales (Child Interference Subscale and Family Interference Subscale). Higher scores are indicative of greater interference of anxiety symptoms in the life of the children and the family.
Changes of children's psychological flexibility | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by The Avoidance and Fusion Questionnaire - Youth (AFQ-Y). AFQ-Y assess children's psychological inflexibility, namely children's experiential avoidance and cognitive fusion. Higher scores are indicative of higher levels of children's psychological inflexibility.
Changes of children's behavioral avoidance | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Child- and Parent-Report Measures of Behavioral Avoidance Related to Childhood Anxiety Disorders (CAMS and CAMP). Higher scores are indicative of higher levels of children's behavioral avoidance.
Changes of children's negative affect | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Positive and Negative Affect for Children (PANAS-C). PANAS-C is composed by two independent subscales: Positive Affect and Negative Affect. Higher scores are indicative of higher levels of children's positive and negative affect, respectively.
Changes of children's negative emotionality | Baseline, Póst-treatment (15 weeks)
  Measured by School-Age Temperament Inventory (SATI). It is composed by five dimensions: negative emotionality, inhibition, adaptability, activity, and persistence. Only the subscale of negative emotionality is used in this study. Higher scores are indicative of higher levels of negative emotionality.
Changes of children's anxiety sensitivity | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Children's Anxiety Sensitivity Inventory-Revised (CASI-R). Higher scores are indicative of higher levels of anxiety sensitivity.
Changes of children's tolerance of negative emotions | Baseline, Mid-treatment (7 weeks), Póst treatment (15 weeks), Follow-up 3 months
  Measured by Distress Tolerance Scale (DTS). Higher scores are indicative of lower levels of tolerance to feel negative emotions.
Changes of children's mindfulness skills | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by The Child and Adolescent Mindfulness Measure (CAMM). Higher scores are indicative of higher levels of children's mindfulness skills.
Changes of children's negative cognitive error | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Children's Negative Cognitive Error Questionnaire (CNCEQ). It assesses four types of cognitive errors derived theoretically: catastrophizing, overgeneralization, personalizing, and selective abstraction. CNCEQ yields a Total Score for each type of cognitive error, a Total Score for areas of content (social, academic, Atlético) and a Total Score for cognitive errors. Higher values correspond to more cognitive errors.
Changes of children's emotional expression and emotion awareness | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Emotional Expression Scale for Children (EESC). Higher scores are indicative of higher levels of difficulties in children's emotional expression and emotion awareness.
Changes of parent's anxiety and depression | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks)
  Measured by Hospital Anxiety and Depression Scale (HADS). Higher scores are indicative of higher levels of anxiety and depression.
Changes of parental anxiety, parental overprotection and parental support of children's coping behaviors | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Parental anxiety and overprotection scale (PAOS). Higher scores are indicative of higher levels of parental anxiety, parental overprotection and parental support of children's coping behaviors.
Changes of parental neuroticism | Baseline, Póst-treatment (15 weeks)
  Measured by NEO Five-Factor Inventory (NEO-FFI). It assesses the five traits of personality defined in the Five Factor Theory of Personality: Openness, Conscientiousness, Extraversion, Agreeableness and Neuroticism. In the present study only Neuroticism subscale was used. Higher scores are indicative of higher levels of neuroticism.
Changes of parental inconsistency and permissiveness | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Parenting Styles & Dimensions Questionnaire. Only the permissiveness subscale was used with higher scores being indicative of higher levels of parental inconsistency and permissiveness.
Changes of parental criticism | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by EMBU-P (egna minnen beträffande uppfostran). It assesses four dimensions: emotional support, rejection, control attempt and sibling preference. In this study, only the rejection subscale was used, which assesses parental rejection and criticism. Higher scores indicate higher levels of rejection and parental criticism.
Changes of shaping of negative emotions | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by The Parent Emotion Regulation Scale (PERS). It assesses four dimensions: parents' orientation to the child's emotions, parents' avoidance of the child's emotions, parents' lack of emotional control and parents' acceptance of the child's and their own emotions. In the present study only parents' lack of emotional control scale was used. This subscale assesses the lack of ability to modulate their own negative emotions in the presence of the child. Higher scores are indicative of higher levels of shaping of negative emotions.
Changes of mindfulness in parenting | Baseline, Mid-treatment (7 weeks), Póst-treatment (15 weeks), Follow-up 3 months
  Measured by Interpersonal Mindfulness in Parenting Scale (IMP). Higher scores are indicative of higher levels of mindfulness in parenting.

OTHER OUTCOMES:
Feasibility of the program by adherence and dropout rate | Póst-treatment (15 weeks)
  Measured through the number of completers and users that dropped out from the intervention before completing it and through the involvement of the participants in the homework (through a record made at each session).
Acceptability of the program | Póst-treatment (15 weeks)
  Measured through specific questions (developed by the researchers) to assess acceptability of the program and to assess satisfaction for each session and for the global intervention - for parents and children; Measured by Parent Motivation Inventory - PMI (to measure parent motivation to participate in treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Brígida Caiado, MsC, Principal Investigator — Faculty of Psychology and Education Sciences, University of Coimbra
Locations (1):
- Faculty of Psychology and Education Sciences, University of Coimbra, Coimbra, Coimbra, Portugal, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Caiado B, Gois A, Pereira B, Canavarro MC, Moreira H. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Children (UP-C) in Portugal: Feasibility Study Results. Int J Environ Res Public Health. 2022 Feb 4;19(3):1782. doi: 10.3390/ijerph19031782. PMID 35162806
- See also: Project webiste — http://protocolounificadoc.wixsite.com/home
- See also: Project facebook — http://www.facebook.com/detetivesemocoesprotocolounificadocriancas